CLINICAL TRIAL: NCT02079519
Title: Bevacizumab as Treatment for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of Avastin (Bevacizumab) in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued prematurely by the sponsor due to a lack of recruitment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18704
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bevacizumab

ARMS (1):
- Bevacizumab 5 mg/kg (Experimental): Participants received bevacizumab 5 mg/kg intravenously every 2 weeks for 6 months until disease progression or termination of the study. Participants showing a continuous benefit of therapy could receive treatment for a maximum of 12 months.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was provided as a concentrate in vials.
  Other Names: Avastin; RO 487-6646

SUMMARY:
This study evaluated the efficacy and safety of Avastin (bevacizumab, 5 mg/kg intravenously every 2 weeks) in patients with multiple myeloma, relapsed/refractory after at least 2 lines of prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 19-75 years of age
* Multiple myeloma.
* Progressive disease after at least 2 lines of prior therapy.

Exclusion Criteria:

* Non-secretory myeloma.
* History of malignancy, other than squamous cell cancer, basal cell cancer, or cancer in situ of the cervix within the last 5 years.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start.
* Clinically significant cardiac disease.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (2):
- Austria (2):
  - Salzburg
  - Vienna

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab 5 mg/kg
Started | 10
Completed | 0
Not Completed | 10
Not completed — Disease Progression | 9
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants who received at least 1 dose of study drug.
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response or a Partial Response
Description: A complete response was defined as the disappearance of the original monoclonal protein from the blood and urine on at least 2 determinations 6 weeks apart; < 5% plasma cells in the bone marrow on at least 2 determinations 6 weeks apart; if a skeletal survey is available, no increase in the size or number of lytic bone lesions; and the disappearance of soft tissue plasmacytomas for at least 6 weeks. A partial response was defined as a ≥ 50% reduction of monoclonal protein in the blood on at least 2 determinations 6 weeks apart; if present, reduction in 24-hour urinary light chain excretion by either ≥ 90% or to < 200 mg for at least 2 determinations 6 weeks apart; ≥ 50% reduction in the size of tissue plasmacytomas for at least 6 weeks; and if a skeletal survey is available, no increase in the size or number of lytic bone lesions.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Intent-to-treat population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 10
Percentage of participants | 0.0

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first dose of study drug to disease progression or death due to progression.
Time Frame: Baseline to the end of the study (up to 1 year)
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first dose of study medication until death.
Time Frame: Baseline to the end of the study (up to 1 year)
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Intent-to-treat population: All participants who received at least 1 dose of study drug.
Arm/Group | Bevacizumab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 5 mg/kg (N=10)
General physical health deterioration (General disorders) | 2
Pyrexia (General disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.